CLINICAL TRIAL: NCT04510129
Title: Predicting Immunotherapy Efficacy from Analysis of Pre-treatment Tumor Biopsies
Brief Title: A Multicenter Cancer Biospecimen Collection Study
Status: Recruiting | Type: Observational
Sponsor: Cofactor Genomics, Inc. (Industry)
Collaborators: Curebase Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PREDAPT
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cancer of Head and Neck; Lung Cancer, Nonsmall Cell; Small-cell Lung Cancer; Urothelial Carcinoma; Gastroesophageal Junction Adenocarcinoma; Cervical Cancer; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Cancer; Hepatocellular Carcinoma; Renal Cell Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Transitional Cell; Uterine Cervical Neoplasms; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sections of subjects' pre-immunotherapy-treatment tumor biopsy, already collected as part of standard of care, will be collected as part of this study. Biopsy specimens may be used in subsequent studies for the development and validation of a diagnostic test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (11):
- head and neck squamous cell carcinoma (HNSCC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- non-small-cell lung cancer (NSCLC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- small cell lung cancer (SCLC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- urothelial carcinoma (UCC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- gastric or gastroesophageal junction adenocarcinoma
  Interventions: Diagnostic Test: OncoPrism™ assay
- cervical cancer
  Interventions: Diagnostic Test: OncoPrism™ assay
- esophageal squamous cell carcinoma (ESCC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- triple-negative breast cancer (TNBC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- hepatocellular carcinoma (HCC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- renal cell carcinoma (RCC)
  Interventions: Diagnostic Test: OncoPrism™ assay
- colorectal cancer (CRC)
  Interventions: Diagnostic Test: OncoPrism™ assay

INTERVENTIONS:
Diagnostic Test: OncoPrism™ assay — OncoPrism™ is a new approach to characterizing the immune component of pre-treatment tumor tissue.

SUMMARY:
This study will collect de-identified tumor samples, with correlated clinical/demographic data and tissue histology, from patients selected or scheduled for pre-treatment tumor biopsy or who have had a recent pre-treatment tumor biopsy. These specimens and clinical data may be used in subsequent studies for the development and validation of a diagnostic test.

DETAILED DESCRIPTION:
This study will establish a prospective cohort of pre-treatment tumor specimens with correlated de-identified clinical and demographic data and tissue histology from cancer patients who are undergoing treatment with PD-1/PD-L1 inhibitors. Patients who have undergone pre-anti-PD-1/PD-L1-treatment tumor biopsy or who are scheduled for tumor biopsy prior to anti-PD-1/PD-L1 treatment will be enrolled.

The study will not require a study-specific tumor biopsy; any biopsies taken prior to treatment as part of standard of care are eligible for this study. Biopsies must not have been taken after immunotherapy treatment began.

Participants will be asked to provide their consent for the potential use of their biospecimens in subsequent studies for the development and validation of a diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a disease of interest. Specifically, subject must have one of:

   1. head and neck squamous cell carcinoma (HNSCC)
   2. non-small-cell lung cancer (NSCLC)
   3. small cell lung cancer (SCLC)
   4. urothelial carcinoma (UCC)
   5. gastric or gastroesophageal junction adenocarcinoma
   6. cervical cancer
   7. esophageal squamous cell carcinoma (ESCC)
   8. triple-negative breast cancer (TNBC)
   9. hepatocellular carcinoma (HCC)
   10. renal cell carcinoma (RCC)
   11. colorectal cancer (CRC)
2. Subject must have received, or be scheduled to receive, at least one dose of anti-PD-1/PD-L1 immunotherapy for treatment of their cancer.
3. Subject must have had, or will have, a tumor biopsy prior to treatment with anti-PD-1/PD-L1 immunotherapy.
4. Subject must have undergone, or will undergo, medical imaging (e.g. CT or MRI) of the tumor prior to treatment with anti-PD-1/PD-L1 immunotherapy.
5. Willing to provide electronic informed consent per IRB-approved protocol.
6. Able to speak, read, and comprehend English fluently.
7. Subject is 18 years of age or older.
8. Subjects must have sufficient tissue available to fulfill the specimen requirements of the study.

Exclusion Criteria:

1. Inability or unwillingness to provide informed consent.
2. Subject who does/did not have one of the cancers listed above (other histologies).
3. Subject has already participated in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone pre-anti-PD-1/PD-L1-treatment tumor biopsy or who are scheduled for tumor biopsy prior to anti-PD-1/PD-L1 treatment will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
PD-L1/PD-1 inhibitor response | 6 months
  No response to treatment with PD-L1/PD-1 inhibitor and response to treatment with PD-L1/PD-1 inhibitor.

CONTACTS AND LOCATIONS:
Overall Officials: Jarret Glasscock, Study Director — Cofactor Genomics
Locations (1):
- Curebase, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flanagan KC, Earls J, Hiken J, Wellinghoff RL, Ponder MM, McLeod HL, Westra WH, Vavinskaya V, Sutton L, Deichaite I, Macdonald OK, Welaya K, Wade J 3rd, Azzi G, Pippas AW, Slim J, Bank B, Sui X, Kossman SE, Shenkenberg TD, Alexander WL, Price KA, Ley J, Messina DN, Glasscock JI, Colevas AD, Cohen EEW, Adkins D, Duncavage EJ. Multicenter validation of an RNA-based assay to predict anti-PD-1 disease control in patients with recurrent or metastatic head and neck squamous cell carcinoma: the PREDAPT study. J Immunother Cancer. 2024 Nov 3;12(11):e009573. doi: 10.1136/jitc-2024-009573. PMID 39489541
- See also: Sponsor Website — https://cofactorgenomics.com/